CLINICAL TRIAL: NCT04095182
Title: A Dose Randomized, Double-blind, Placebo Controlled, Single and Multiple Dosing, Dose-escalation Phase I Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetic Characteristics of Zebinix (Eslicarbazepine Acetate) After Oral Administration in Healthy Korean and Caucasian Adult Subjects
Brief Title: Clinical Trial for Zebinix (Eslicarbazepine Acetate) in Healthy Korean and Caucasian Adult
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Whanin Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: WID-ESL18-P1
Record Dates: First submitted 2019-09-15; First posted 2019-09-19 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Partial-onset Seizures With or Without Secondary Generalisation
MeSH Terms: interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Zebinix 400mg (Experimental)
  Interventions: Drug: Zebinix 400mg
- Placebo for Zebinix 400mg (Placebo Comparator)
  Interventions: Drug: Placebo for Zebinix 400mg
- Zebinix 800mg (Experimental)
  Interventions: Drug: Zebinix 800mg
- Placebo for Zebinix 800mg (Placebo Comparator)
  Interventions: Drug: Placebo for Zebinix 800mg
- Zebinix 1600mg (Experimental)
  Interventions: Drug: Zebinix 1600mg
- Placebo for Zebinix 1600mg (Placebo Comparator)
  Interventions: Drug: Placebo for Zebinix 1600mg

INTERVENTIONS:
Drug: Zebinix 400mg — Zebinix 400mg group is administered with two Zebinix 200mg tablets per day. (Single dose: Day 1, Multiple dose: Day5~11)
  Arms: Zebinix 400mg
Drug: Placebo for Zebinix 400mg — Placebo for Zebinix 400mg group is administered with two placebo for Zebinix 200mg tablets per day.
  (Single dose: Day 1, Multiple dose: Day5~11)
  Arms: Placebo for Zebinix 400mg
Drug: Zebinix 800mg — Zebinix 800mg group is administered with a Zebinix 800mg tablet per day. (Single dose: Day 1, Multiple dose: Day5~11)
  Arms: Zebinix 800mg
Drug: Placebo for Zebinix 800mg — Placebo for Zebinix 800mg group is administered with a placebo for Zebinix 800mg tablets per day.
  (Single dose: Day 1, Multiple dose: Day5~11)
  Arms: Placebo for Zebinix 800mg
Drug: Zebinix 1600mg — Zebinix 1600mg group is administered with two Zebinix 800mg tablets per day. (Single dose: Day 1, Multiple dose: Day5~11)
  Arms: Zebinix 1600mg
Drug: Placebo for Zebinix 1600mg — Placebo for Zebinix 1600mg group is administered with two placebo for Zebinix 800mg tablets per day.
  (Single dose: Day 1, Multiple dose: Day5~11)
  Arms: Placebo for Zebinix 1600mg

SUMMARY:
A dose randomized, double-blind, placebo controlled, single and multiple dosing, dose-escalation phase I clinical trial to investigate the safety, tolerability and pharmacokinetic characteristics of Zebinix (Eslicarbazepine acetate) after oral administration in healthy Korean and Caucasian adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged 19-45 years at screening
* Subjects who weigh more than 50kg with a body mass index(BMI) of 18.0~28.0 kg/m2 at screening
* Subjects who are fully understood after being given the detailed explanation of this clinical trial and willing to give written informed consent for participation prior to the screening test
* Subjects who are qualified to participate in this clinical trial through the physical examination, clinical laboratory test and interview by the investigators

Exclusion Criteria:

* Clinically significant presence or treatment history of cardiovascular, hepatic, renal, gastrointestinal, respiratory, neurological, hematological, endocrine, psychiatric
* Clinically significant surgical history
* Clinically significant family history
* Clinically significant atopic syndrome
* History of hypersensitivity or clinically significant hypersensitivity to drug including carbamazepine and related compounds
* History of alcoholism or drug abuse or show a positive response to an abuse drug in the urine drug screening test
* Consistently consume alcohol or cannot stop drinking during the clinical trial
* Smoker
* Significant infection or inflammatory finding at screening visit
* History of gastrointestinal disorders or surgery which may have an effect on the safety and pharmacokinetic evaluation of the investigational products (except for simple appendectomy and herniotomy)
* Have used prescription drugs or herbal medication within 2 weeks of initial administration or who have used over the counter(OTC), health functional food or vitamins within 1 week of initial administration (but, if the other conditions are suitable according to the judgment of the investigator, they can participate in the clinical trial), or subjects who have expected to take it
* Have participated in any clinical trial (or bioequivalence study) and administered any investigational product within 6 months
* Positive for HbsAg, anti-HCV and HIV antigen-antibody reaction tests at screening
* Have donated any whole blood or apheresis or received blood transfusion within 3 months of initial administration of this clinical trial
* Have dietary restrictions or cannot take the food provided by the institution
* Cannot communicate reliably with the investigator
* Subjects who are determined by the investigator to be ineligible for participation in this clinical trial due to clinical laboratory test results or other reasons

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Time of maximum observed drug concentration (Tmax) | 'Day 1' 0(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose, 'Day 6~Day 11' 0 hour(pre-dose), 'Day 11' 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose
Maximum observed plasma drug concentration (Cmax) | 'Day 1' 0(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose, 'Day 6~Day 11' 0 hour(pre-dose), 'Day 11' 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose
Area under the plasma concentration time-curve (AUC) | 'Day 1' 0(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose, 'Day 6~Day 11' 0 hour(pre-dose), 'Day 11' 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose
Apparent terminal elimination half-life (t1/2) | 'Day 1' 0(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose, 'Day 6~Day 11' 0 hour(pre-dose), 'Day 11' 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose
Peak trough fluctuation (PTF) | 'Day 1' 0(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose, 'Day 6~Day 11' 0 hour(pre-dose), 'Day 11' 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose
Accumulation ratio (R) | 'Day 1' 0(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose, 'Day 6~Day 11' 0 hour(pre-dose), 'Day 11' 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose
Metabolic ratio | 'Day 1' 0(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose, 'Day 6~Day 11' 0 hour(pre-dose), 'Day 11' 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 hour post-dose

SECONDARY OUTCOMES:
Adverse event | Day -1 ~ Day 15

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Whan In Pharm., Seoul, South Korea